CLINICAL TRIAL: NCT02101879
Title: Cardiotoxicity in Metastatic Her 2 Positive Patients Treated With First Line Trastuzumab, Pertuzumab and Taxanes Based Regimen
Brief Title: Cardiotoxicity in Metastatic Her 2 Positive Patients Treated With Trastuzumab ,Pertuzumab and Taxanes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiotoxicity
Record Dates: First submitted 2014-03-05; First posted 2014-04-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Cardiotoxicity.; Anti Her2 Therapy.; Metastatic Breast Cancer
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood samples for TNI & BNP will be sent before every cycle for the first 5 cycles of treatment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer Her2 positive: Trastuzumab & Pertuzumab & Taxanes

SUMMARY:
Approximately 15-25% of all breast cancers are human epidermal growth factor receptor 2 (HER2) positive and it has been well known that HER2 overexpression is associated with more aggressive phenotype and poor prognosis with resistance to certain chemotherapeutic agents.

Trastuzumab administration as an adjuvant and in metastatic HER2 positive breast cancer is associated with both symptomatic and asymptomatic cardiotoxicity. The incidence of trastuzumab-mediated cardiotoxicity were 27% with antracycline combination and 13% when it was administered with paclitaxel .

Pertuzumab, a recombinant humanized monoclonal antibody binding to the HER2 dimerization domain, prevents dimerization of HER2 with other HER receptors (HER3,HER1, and HER4) especially with HER3. Blocking HER2-HER3 dimerization is postulated to be the most clinically relevant action of pertuzumab and this can effectively block her2-mediated cell signaling.

Pertuzumab is indicated in combination with trastuzumab and docetaxel for the treatment of patients with HER2-positive metastatic breast cancer who have not received prior anti-HER2 therapy or chemotherapy for metastatic disease.

Treatment of breast cancer with pertuzumab plus trastuzumab plus docetaxel as first line treatment until disease progression might be complicated by cardiotoxicity in up to 14.5% of the Patients.

Cardinale et al showed that troponin I (TNI) positive identifies trastuzumab-treated patients who are at risk for cardiotoxicity and are unlikely to recover from cardiac dysfunction despite HF therapy.

There is very little data about the reversibility and identification of patients at risk for cardiotoxicity of the pertuzumab plus trastuzumab plus docetaxel regimen and of those who will not recover from cardiac dysfunction,this information is crucial. The usefulness of troponin I (TNI) and Brain natriuretic peptide (BNP) in the identification of patients at risk for PT cardiotoxicity and in the prediction of LVEF recovery has never been investigated.

based on this background , this study aim is to evaluate the cardiotoxicity of pertuzumab plus trastuzumab plus docetaxel regimen and the application of troponin I (TNI) and Brain natriuretic peptide (BNP) in this setting.

DETAILED DESCRIPTION:
Breast cancer is the leading cancer in women in Israel with 4000 new cases every year.

Approximately 15-25% of all breast cancers are human epidermal growth factor receptor 2 (HER2) positive and it has been well known that HER2 overexpression is associated with more aggressive phenotype and poor prognosis with resistance to certain chemotherapeutic agents.

Trastuzumab, an anti-HER2 humanized monoclonal antibody, is the standard treatment for both early and metastatic HER2-positive breast cancer. In addition to other chemotherapeutic agents, trastuzumab significantly improves response rate and survival in HER2-positive early and metastatic breast cancer. Although it is well known that trastuzumab therapy is closely associated with both symptomatic and asymptomatic cardiotoxicity.

Addition of trastuzumab to chemotherapy significantly improved response rate, time to disease progression and reduction of death compared to chemotherapy alone in HER2-positive metastatic breast cancer (MBC). Thus, anti-HER2 treatment is a standard therapeutic approach for HER2-positive MBC patients with visceral crisis. Trastuzumab administration as an adjuvant and in metastatic HER2 positive breast cancer is associated with both symptomatic and asymptomatic cardiotoxicity. The incidence of trastuzumab-mediated cardiotoxicity were 27% with antracycline combination and 13% when it was administered with paclitaxel .

Pertuzumab, a recombinant humanized monoclonal antibody binding to the HER2 dimerization domain, prevents dimerization of HER2 with other HER receptors (HER3,HER1, and HER4) especially with HER3. Pertuzumab differs from trastuzumab in the epitope binding regions of the light chain; pertuzumab binds to domain 2 ofHER2 essential for dimerization, whereas trastuzumab binds to domain 4 of HER2. Blocking HER2-HER3 dimerization is postulated to be the most clinically relevant action of pertuzumab and this can effectively block her2-mediated cell signaling.

Pertuzumab is indicated in combination with trastuzumab and docetaxel for the treatment of patients with HER2-positive metastatic breast cancer who have not received prior anti-HER2 therapy or chemotherapy for metastatic disease.

The randomized, double-blind, placebo controlled,phase III CLEOPATRA (the CLinical Evaluation OfPertuzumab And Trastuzumab) study involved 808 patients with HER2-positive MBC who had not received prior chemotherapy or biologic therapy, who were randomized to placebo plus trastuzumab plus docetaxel or pertuzumab plus trastuzumab plus docetaxel as first line treatment until disease progression. No additional cardiotoxicity was observed when adding pertuzumab compared to placebo. The incidence of any cardiac disorder as assessed by the investigators was similar in the placebo (16.4%) and pertuzumab (14.5%) arms. Left ventricular systolic dysfunction (LVSD) was observed in 8.3% and 4.4% of placebo and pertuzumab patients, respectively. Left ventricular systolic dysfunction of grade III or higher was reported in 7 (1.8%) patients in the placebo arm and 4 (1.0%) in the pertuzumab arm.

Treatment of breast cancer with pertuzumab plus trastuzumab plus docetaxel as first line treatment until disease progression might be complicated by cardiotoxicity in up to 14.5% of the Patients.

Cardinale et al showed that troponin I (TNI) positive identifies trastuzumab-treated patients who are at risk for cardiotoxicity and are unlikely to recover from cardiac dysfunction despite HF therapy.

There is very little data about the reversibility and identification of patients at risk for cardiotoxicity of the pertuzumab plus trastuzumab plus docetaxel regimen and of those who will not recover from cardiac dysfunction,this information is crucial. The usefulness of troponin I (TNI) and Brain natriuretic peptide (BNP) in the identification of patients at risk for PT cardiotoxicity and in the prediction of LVEF recovery has never been investigated.

based on this background , this study aim is to evaluate the cardiotoxicity of pertuzumab plus trastuzumab plus docetaxel regimen and the application of troponin I (TNI) and Brain natriuretic peptide (BNP) in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Breast Cancer patients with Her2 Positive Disease.
* No prior treatment

Exclusion Criteria:

* LEVF less than 50%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Metastatic Breast Cancer Her2 Positive
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
To assesses blood levels of TNI and BNP during the first four cycles Trastuzumab&Pertuzumab and Taxanes treatment | The patients will be followed until the end of therapy (an expected average of 18 months).
  Prior to every treatment cycle, blood samples will be taken for TNI & BNP. Patients with elevated levels will be sent for LEVF evaluation. In cases with LEVF reduction of 15% or more from the baseline or LEVF less than 50% will be sent for Cardiological consult in order to consider ACEI or BB treatment
To evaluate the correlation between elevated TNI&BNP and decline of LVEF on echocardiography until end of treatment. | The patients will be followed until the end of therapy (an expected average of 18 months).
  Prior to every treatment cycle, blood samples will be taken for TNI & BNP. Patients with elevated levels will be sent for LEVF evaluation. In cases with LEVF reduction of 15% or more from the baseline or LEVF less than 50% will be sent for Cardiological consult in order to consider ACEI or BB treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam MC, Haifa, Israel